CLINICAL TRIAL: NCT07355192
Title: Group Singing (Hybrid Format) or Solo Singing in Older Adults With Coronary Artery Disease: A Feasibility Study
Brief Title: Hybrid Group Singing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jacquelyn Kulinski, Professor of Medicine/Cardiology, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 00056785
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Elderly
Keywords: group singing; individual singing
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Parallel with baseline hybrid group randomized design
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group singing (hybrid format) (Active Comparator): Group singing sessions are a hybrid of in-person and virtual participation with in-person participation encouraged. Intake forms will be used to assess musical preference, prior music experience, and pertinent medical conditions to consider. Songs will be selected based on music preference of the subjects. At the start of each session, the music therapist will review the importance of singing and lead the group in taking deep breaths together. Throughout sessions, the therapist will encourage subjects to sing as much as possible, explaining that it's not about how they sound but how they feel. Initially, the group singing format will be 40 minutes of singing (includes a vocal warm-up), three times weekly, for a total of 12 weeks. The total singing time is the same as in the solo singing video arm. Based on focus group feedback, the formats could change. However, we will aim to keep total singing time the same (i.e., 120 minutes of singing per week).
  Interventions: Behavioral: group singing (hybrid format)
- individual sing-along video series (Active Comparator): Participants in this arm watch and sing to an online video series independently. The video series is created by a professor of voice with older students in the videos. We plan to use REDCap to deliver the assigned videos at set times and frequencies and display the videos in an embedded audio player for the subjects. Use of REDCap will allow us to track when subjects are watching the videos with reminders sent up to five times. We will also include 2 questions at the end on how much they enjoyed the video (scale 1-10) and how much of the 40 minutes were sung. Inserting questions at the end confirms that participants likely viewed the entire video.
  Interventions: Behavioral: instructional sing-along video series

INTERVENTIONS:
Behavioral: group singing (hybrid format) — 12-weeks of group singing, combination of in-person and virtual sessions, 3 times weekly
  Arms: group singing (hybrid format)
Behavioral: instructional sing-along video series — 12-week solo singing video series done independently, 3 times weekly
  Arms: individual sing-along video series

SUMMARY:
The overall objective of the planned future clinical trial is to test the investigator's central hypothesis that habitual singing over several weeks, similar to habitual exercise, will lead to sustained and favorable vascular adaptation, thereby lowering cardiovascular disease (CVD) risk. The overall objective of this study is to refine and protocolize the singing interventions and test the feasibility of the future trial design. The investigative team has previously studied solo singing. Collective singing, as in a choir or small group, is associated with a positive sense of social inclusion, well-being, and improved mood, including in older adults.

DETAILED DESCRIPTION:
The investigator previously studied 65 subjects (mean age 68±7, 40% women) with known CAD in a randomized, control cross-over clinical trial of singing interventions: (1) a 30-minute period of guided singing from an in-person coach (music therapist), (2) a 30-minute period of singing along to an instructional video created by and including a professor of voice and 'inexperienced, older singing student,' and (3) a 'rest' control during which subjects underwent a brief hearing test. Fifty-four percent reported a physical or orthopedic limitation. The primary outcome was vascular endothelial function. There was statistically significant improvement in microvascular endothelial function, as measured by the Framingham reactive hyperemia index (fRHI), after 30 minutes of singing in the instructional video arm (30.9%, p=0.007) compared to the rest control. The observed change in fRHI in the prior clinical trial translates into a ~25% reduction in CVD risk, which is comparable to traditional cardiac rehabilitation program participation. There was no improvement in macrovascular function, as assessed by brachial artery flow-mediated dilation. The visit with the music therapist coach did not reach statistical significance. Unfortunately, this may have been related to disruption of the in-person coach visits during the COVID pandemic, where the investigator continued the clinical trial but moved to a virtual interaction for the one-on-one coach visits (n=20 out of 65 subjects).

Why should group singing be considered? Collective singing, as in a choir or small group, is associated with a positive sense of social inclusion, well-being, and improved mood (less anxiety and depression), including in older adults and may be less anxiety-provoking than one-on-one singing. From a healthcare systems standpoint, group singing would be more efficient and cost-saving (lower per-person cost than individual singing therapy), which has been shown for other treatments without compromising efficacy. With a longer intervention planned for 12 weeks, there will be ample opportunity for the therapeutic relationship between patients and music therapist. The investigator needs to show that this acute, beneficial vascular adaptation is sustained after habitual singing over several weeks, thereby lowering future CVD risk. Before the investigator can execute a large-scale efficacy trial, the study team needs to determine the most acceptable frequency, duration, and delivery format (in-person and/or virtual) that is feasible and tailored to the target population. This study will help the investigator and team protocolize the group singing and video interventions, execute a feasibility trial on a smaller scale, and assess the fidelity of the delivered interventions in preparation for the larger efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* history of coronary artery disease (defined as having at least 1 of the following: myocardial infarction, coronary stent, PCI, CABG, coronary stenosis at least 50%, or coronary artery calcification score at least 300 Agatston units)

Exclusion Criteria:

* Parkinson's disease or tremor
* upper arm fistula
* fingernail onychomycosis
* pregnancy
* current tobacco use
* current illicit drug use
* current excessive alcohol use (defined as more than 14 drinks/week for women, more than 28 drinks/week for men)
* unstable CAD (active symptoms of chest discomfort)
* supplemental oxygen use
* more than mild cognitive impairment (as documented in the medical record by patient's treatment teams)
* inability to follow study procedures
* non-English speaking

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Adherence | 12 weeks
  The mean percent of sessions attended.

SECONDARY OUTCOMES:
Enrollment rate | 12 weeks
  Proportion of subjects who enroll out of all approached, eligible patients and participate in at least one session.
Retention rate | out of 2 study visits (baseline and post-intervention visit after 12 weeks)
  Proportion of enrolled subjects who complete all study visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Bagherimohamadipour M, Hammad M, Visotcky A, Sparapani R, Kulinski J. Effects of singing on vascular health in older adults with coronary artery disease: a randomized, crossover trial. Front Cardiovasc Med. 2025 Apr 28;12:1546462. doi: 10.3389/fcvm.2025.1546462. eCollection 2025. PMID 40357442